CLINICAL TRIAL: NCT03052101
Title: Assessment of Safety of Air Travel in Patients With Pulmonary Langerhans Cell Histiocytosis
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nishant Gupta, MD, MS, Assistant Professor, University of Cincinnati
Other Study IDs: RLDC5714B; U54HL127672 (NIH)
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Langerhans Cell Histiocytosis
Keywords: PLCH; Air travel; pneumothorax; pleurodesis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Pneumothorax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to conduct survey-based assessments for the safety of air travel in patients with pulmonary Langerhans cell histiocytosis (PLCH). The study will enroll patients through the clinic network at Rare Lung Disease Consortium (RLDC) and through the Histiocytosis Association website. Patients will have access to the questionnaire via REDCap (an online data management system) and each patient will be provided with a link to complete the survey. The investigators plan on enrolling approximately 200 patients with PLCH for the purpose of this study. Secondary aims of this study include further characterization of the clinical aspects of disease and to establish a contact registry for these patients, in order to facilitate future studies.

DETAILED DESCRIPTION:
The study will enroll participants through the clinic network at the Rare Lung Disease Consortium (RLDC) and through the Histiocytosis Association websites. Participants will have access to the questionnaire via REDCap (an online data management system) and each participant will be provided a link to complete the survey. In case of lack of internet access or inability to complete the online questionnaire, a paper survey will be mailed out with a pre-paid envelope to return the survey.

Primary Study Objective(s):

To define the risk of pneumothorax associated with air travel in patients with PLCH.

Secondary Study Objective(s):

To establish a contact registry for patients with PLCH to facilitate future trials To assess the rate of pneumothorax recurrence in patients with PLCH To assess the efficacy of pleurodesis in preventing recurrent pneumothoraces among patients with PLCH

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 18 or older
* English literate
* Signed, dated informed consent; either given electronically or via paper form
* Confirmed diagnosis of PLCH based either on characteristic radiologic findings, or histopathological confirmation

Exclusion Criteria:

* Inability, or refusal, to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Pulmonary Langerhans Cell Histiocytosis
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Singla A, Kopras EJ, Gupta N. Spontaneous pneumothorax and air travel in Pulmonary Langerhans cell histiocytosis: A patient survey. Respir Investig. 2019 Nov;57(6):582-589. doi: 10.1016/j.resinv.2019.07.004. Epub 2019 Sep 26. PMID 31563637
- See also: Link to completing the online study questionnaire — https://redcap.research.cchmc.org/surveys/?s=C7EY4WNPEY

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort: Self-reported PLCH participants who completed an online survey.
Period: Overall Study
Arm/Group | Cohort
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort
Number analyzed (Participants) | 94
Age, Continuous [Mean (Full Range); unit: years] | 47 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 90
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PLCH Who Experienced Spontaneous Pneumothorax During or Within 24 Hours Following Air Travel
Description: The investigators will measure the number of pneumothoraces that occur either during air travel, or within 24 hours of air travel among patients with pulmonary Langerhans cell histiocytosis. The incidence of air travel related pneumothorax will be calculated by dividing the number of pneumothoraces to the total number of flights undertaken by the entire cohort.
Time Frame: During air travel or within 24 hours following air travel
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 94
Participants | 2

2. Secondary Outcome: Number of Patients With Pulmonary Langerhans Cell Histiocytosis Who Experienced a Spontaneous Pneumothorax
Description: The investigators will catalogue the number of spontaneous pneumothoraces experienced by patients with pulmonary Langerhans cell histiocytosis.
Time Frame: 2 years and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 94
Participants | 22

3. Secondary Outcome: Number of Patients With Pulmonary Langerhans Cell Histiocytosis Who Experienced Recurrent Pneumothorax
Description: The investigators will measure the number of participants who experience a recurrent spontaneous pneumothorax.
Time Frame: 2 years and 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort: Self-reported PLCH participants who experienced recurrent spontaneous pneumothorax.
Arm/Group | Cohort
Number analyzed (Participants) | 22
Participants | 14

ADVERSE EVENTS:
Time Frame: This was a cross-sectional survey, filled out online. The only risk was potential data breech. All-cause mortality, serious adverse events and other adverse events were not collected as part of this study.
Description: This was a cross-sectional survey, filled out online. The only risk was potential data breech. All-cause mortality, serious adverse events and other adverse events were not collected as part of this study.
Arm/Group | Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT03052101/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT03052101/ICF_001.pdf